CLINICAL TRIAL: NCT04105296
Title: Epidural Stimulation for Locomotion After Spinal Cord Injury
Brief Title: Epidural Stimulation After Spinal Cord Injury
Acronym: ESL-SCI
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGuire Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2501
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- EKSO+ES (Experimental): 6 months of exoskeleton training with spinal cord epidural stimulation.
  Interventions: Device: EKSO+ES

INTERVENTIONS:
Device: EKSO+ES — 6 months of exoskeleton training with epidural stimulation.

SUMMARY:
The purpose of the current study is to determine the effects of applying epidural stimulation (ES) on motor control recovery in Veterans with SCI. The intervention will be accompanied with the use of a powered exoskeleton (EKSO®) for 6 months to facilitate standing and to produce step-like movement in persons with chronic motor complete (AIS A or B) SCI and level of injury below C5 . Walking speed, distance, muscle activation pattern as measured by surface EMG and walking parameters including stand-up time, walking time, distance will be considered primary outcome variables. Cardiovascular performance, as measured by resting blood pressure and heart rate, peak oxygen consumption during walking, energy expenditure, whole and regional body composition assessments will also be measured. The effects of training (ES+EKSO) on , and speed of walking will also be evaluated.

DETAILED DESCRIPTION:
Five veterans with chronic motor complete SCI (AIS A or B) will be recruited to participate in the current trial. The primary objective is to determine how implantation of an epidural stimulator can help to control movement in the leg muscles to stand and perform stepping. Participants will be trained using a robotic suit and parallel bars. The procedure of using epidural stimulation with the robotic suit is experimental. The participant will be scheduled to perform temporary implantation followed by permanent implantation. Seven days later, two 8-electrode arrays of Vectris lead will be implanted in an operating room. The research team will be responsible for helping the participants to trigger the paralyzed muscles from supine and sitting using for 5 days per week. Participants would be required to come for study visits twice daily for 2 hours per day. Each visit will last approximately 1 hour in the morning and 1 hour in the evening. During these visits, participants will practice walking with a robotic suit for 30-60 minutes followed by overground walking between parallel bars, or with a walker or crutches.

ELIGIBILITY:
Inclusion Criteria:

1. A written clearance by the medical doctor to ensure that the participant is safely able to engage in the program.
2. Participants who require assistance with activities of daily living, must have a caregiver or companion with them throughout their participation in the study.
3. Participants will have to be 2 years post-injury with any level of injury below C5 and using wheelchair as the primary mode of mobility. The study is primarily exploratory, and all participants will be between 18-70 years old with SCI.
4. Hip width (distance between two greater trochanters), upper leg length (greater trochanter to the lateral aspect of joint line of the knee joint) and lower leg length (lateral aspect of joint line of the knee joint to the bottom of the foot) that can fit the robotic suit.

Exclusion Criteria:

1. Unhealed fracture in either lower or upper extremities
2. Severe scoliosis, hip knee ROM or flexion knee contractures preventing positioning in an exoskeleton or plantarflexion deformity greater than 20 degrees.
3. High resting blood pressure greater than 140/80 mmHg and or sudden hypotension upon standing as characterized by drop in blood pressure by 20 mmHg especially in persons with tetraplegia.
4. Other medical conditions including cardiovascular disease, uncontrolled type II DM, uncontrolled hypertension, and those on insulin, pressures sores stage 3 or greater, or symptomatic urinary tract infection.
5. Unable to fit in the device for any reason.
6. Taking anti-coagulants or anti-platelet agents, including aspirin if unable to be off this medication for medical reasons.
7. Implanted pacemakers and/or implanted defibrillator devices.
8. Any condition that, in the judgment of the principal investigator or medical provider, precludes safe participation in the study and/or increases the risk of infection.
9. Dual Energy X-ray Absorptiometry (DXA) T-Score less than -2.5. Scans done will include total body, dual hips and knees.
10. Functional upper and lower extremity range of motion (ROM), strength, spasticity and skin integrity will also have assessed prior to enrollment in the program. The Modified Ashworth Scale will be used to ensure safety of the participants prior to engagement in the rehabilitation program. Participants with severe spasticity or limited ROM will be excluded in the trial. This will be done based on the manufacture's recommendation.
11. Other exclusion criteria may include the followings

    * subjects with uncontrolled autonomic dysreflexia
    * subjects with concurrent severe neurological injuries other than SCI: MS, CP, TBI, stroke;
    * subjects with unresolved deep vein thrombosis (DVT);
    * subjects with prosthetic lower limbs;
    * subjects with psychiatric or cognitive impairments which will interfere with proper operation of both the spinal cord stimulator as well as the exoskeleton;
    * subjects with an unhealed spinal fracture or unstable spine; and
    * subjects with known cardiac pathology which precludes safe participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Six minute-walk and 10-meter walk distance Tests | 6 months
  Walking distance and speed will also be determined
Surface electromyography of 6 different muscle groups | 6 months
  The EMG activity from 6 major leg muscles will be measured during locomotion

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure | 6 months
  During sitting, standing and walking
Oxygen uptake using Portable Indirect Calorimetry | 6 months
  During sitting, standing and walking
Body composition assessment of fat mass and fat-free mass using dual energy x-ray absorptiometry (DXA) | 6 months
  Before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Gorgey, PhD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be available in the form of published case reports as well as scientific presentations in national and international meetings.